CLINICAL TRIAL: NCT06832371
Title: Evaluation of the Effect of Lomitapide Treatment on Major Adverse Cardiovascular Events (MACE) in Patients With Homozygous Familial Hypercholesterolemia: A Multicenter, Retrospective and Prospective Observational Study
Brief Title: Evaluation of the Effect of Lomitapide Treatment on Major Adverse Cardiovascular Events (MACE) in Patients With Homozygous Familial Hypercholesterolemia
Acronym: LILITH
Status: Recruiting | Type: Observational
Sponsor: Fondazione SISA (Societa Italiana per lo Studio della Arteriosclerosi) (Other)
Collaborators: Amryt Pharmaceuticals DAC (Unknown); Clinical Trial Consulting (Unknown); CMV-Stat S.r.l. (Unknown)
Responsible Party: Sponsor
Other Study IDs: LILITH
Record Dates: First submitted 2025-02-10; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Homozygous Familial Hypercholesterolemia (HoFH); Major Adverse Cardiovascular Events (MACE); Dyslipidemia
Keywords: Lomitapide; Hypercholesterolemia; Cardiovascular Disease; LDL Cholesterol; Lipid-Lowering Therapy; Lipid Metabolism Disorders; Atherosclerosis; Rare Genetic Disorders
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Dyslipidemias; Hypercholesterolemia; Cardiovascular Diseases; Lipid Metabolism Disorders; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples will be collected and retained for lipid profile analysis, liver function tests (ALT, AST, GGT), and other biochemical assessments related to the study objectives. No genetic testing or DNA extraction will be performed on the retained samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HoFH Patients Treated with Lomitapide: This cohort consists of adult patients (≥18 years) diagnosed with Homozygous Familial Hypercholesterolemia (HoFH) who have been treated with lomitapide for at least 12 months. The study will retrospectively analyze the incidence of Major Adverse Cardiovascular Events (MACE) in the three years before lomitapide treatment, and prospectively track MACE incidence during the first three years of lomitapide therapy.

SUMMARY:
This observational, multicenter, retrospective and prospective study aims to evaluate the effect of lomitapide treatment on Major Adverse Cardiovascular Events (MACE) in patients with Homozygous Familial Hypercholesterolemia (HoFH).

HoFH is a rare genetic disorder characterized by extremely high levels of LDL cholesterol (LDL-C), leading to an increased risk of early cardiovascular diseases. Lomitapide is an approved medication that lowers LDL-C levels by inhibiting microsomal triglyceride transfer protein (MTP).

The study will collect data from patients who have been treated with lomitapide for at least 12 months and will compare the incidence of MACE during the first three years of treatment with the three years before treatment initiation. The study includes data collection from multiple lipid centers across Europe.

The primary objective is to assess the impact of lomitapide on MACE, while secondary objectives include evaluating changes in lipid profiles, liver function tests, and lipid-lowering treatments.

DETAILED DESCRIPTION:
This is a multicenter, international, long-term observational study investigating the real-world impact of lomitapide on Major Adverse Cardiovascular Events (MACE) in patients with Homozygous Familial Hypercholesterolemia (HoFH).

Study Design:

Observational, open-label, retrospective and prospective study Data will be collected from >26 lipid centers across Europe Patients will serve as their own control, with comparisons between pre-treatment (3 years before lomitapide) and post-treatment (first 3 years of lomitapide therapy) periods

Study Population:

Approximately 72 adult patients (≥18 years) diagnosed with HoFH Patients must have received lomitapide for at least 12 months Availability of 3 years of pre-treatment clinical records

Objectives:

Primary Objective: Evaluate the incidence of MACE before and after lomitapide treatment

Secondary Objectives: Assess changes in LDL-C, total cholesterol, liver function tests (ALT, AST, GGT), and lipid-lowering therapy usage (e.g., discontinuation of LDL apheresis, addition of PCSK9 inhibitors)

Endpoints:

Primary Endpoint: Change in MACE incidence over the 3-year treatment period

Secondary Endpoints: Changes in lipid levels, liver safety markers, and adherence to treatment protocols

Safety Considerations:

The study follows real-world clinical practice, with monitoring of adverse events, including liver-related safety concerns associated with lomitapide

Data will be collected in an electronic Case Report Form (eCRF) and analyzed following Good Clinical Practice (GCP) guidelines

This study aims to generate real-world evidence on the cardiovascular impact of lomitapide in HoFH patients, addressing an unmet clinical need for data on long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years)
* Clinical or genetic diagnosis of HoFH
* Treated with lomitapide at any dosage
* On treatment with lomitapide for at least 12 months at the time of enrollment
* Availability of 3 years of medical records prior to lomitapide treatment to confirm MACE
* Giving written informed consent

Exclusion Criteria:

* Patients who were prescribed lomitapide outside of the marketing authorization or in contraindicated patients
* Patients receiving lomitapide in clinical trials
* Patients receiving an investigational agent, defined as any drug or biologic agent other than lomitapide that has not received Market Authorization in the country of participation, at the time of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical or genetic diagnosis of homozygous familial hypercholesterolemia (HoFH) who have been treated with lomitapide for at least 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) Before and After Lomitapide Treatment | 3 years before treatment vs. 3 years during treatment
  This measure will assess the incidence of MACE (including myocardial infarction, stroke, cardiovascular death, and hospitalization due to unstable angina) during the first three years of lomitapide treatment compared to the three years prior to treatment initiation.
  Unit of Measure: Number of events per 100 patient-years.

SECONDARY OUTCOMES:
Change in LDL-Cholesterol Levels | Baseline, 1 year, 2 years, 3 years
  This measure will evaluate changes in LDL-C levels. Unit of Measure: mg/dL.
Change in Total Cholesterol, Triglycerides, and HDL-Cholesterol | Baseline, 1 year, 2 years, 3 years
  Assess changes in total cholesterol, triglycerides, and HDL-C at 1, 2, and 3 years after lomitapide treatment initiation.
  Unit of Measure: mg/dL.
Change in Triglyceride Levels | Baseline, 1 year, 2 years, 3 years.
  This measure will evaluate changes in triglyceride levels. Unit of Measure: mg/dL.
Change in HDL-Cholesterol Levels | Baseline, 1 year, 2 years, 3 years
  This measure will evaluate changes in HDL-C levels. Unit of Measure: mg/dL.
Liver Safety Profile - ALT Levels | Baseline, 1 year, 2 years, 3 years.
  This measure will evaluate changes in alanine aminotransferase (ALT) levels. Unit of Measure: U/L.
Liver Safety Profile - AST Levels | Baseline, 1 year, 2 years, 3 years.
  This measure will evaluate changes in aspartate aminotransferase (AST) levels. Unit of Measure: U/L.
Liver Safety Profile - GGT Levels | Baseline, 1 year, 2 years, 3 years.
  This measure will evaluate changes in gamma-glutamyl transferase (GGT) levels. Unit of Measure: U/L.
Lipid-Lowering Therapy Modifications | Baseline, 1 year, 2 years, 3 years.
  This measure will track changes in lipid-lowering therapies, for example the discontinuation of LDL apheresis or the introduction of evinacumab, as described in the study protocol.
  Unit of Measure: Number of patients with therapy modifications.

OTHER OUTCOMES:
Biomarkers of Liver and Vascular Damage | Baseline and after 3 years of lomitapide treatment.
  This measure will evaluate biomarkers of liver and vascular damage, including FIB4, apolipoprotein B, lipoprotein(a), cytokeratin 18 fragment (CK-18F), hematology, and other relevant markers.
  Unit of Measure: Laboratory values in mg/dL or U/L, as applicable.
Presence and Severity of Hepatic Steatosis | After 3 years of lomitapide treatment.
  This measure will assess the presence and severity of hepatic steatosis using liver ultrasound or MRI. Severity will be graded as absent, mild, moderate, or severe.
  Unit of Measure: Qualitative assessment (absent, mild, moderate, severe).
Liver Elastography Parameters | After 3 years of lomitapide treatment.
  This measure will evaluate liver elastography parameters using fibroscan or other methods. Measurements will include liver stiffness (kPa) and controlled attenuation parameter (CAP) values.
  Unit of Measure: kPa (kilopascal) and CAP (dB/m).
Dietary Records | After 3 years of lomitapide treatment.
  This measure will evaluate dietary patterns using a food frequency questionnaire (FFQ) for patients participating in the prospective phase of the study.
  Unit of Measure: Responses to FFQ (categorical and quantitative data).
Adherence to Lipid-Lowering Medications | After 3 years of lomitapide treatment.
  This measure will evaluate adherence to lipid-lowering medications, including lomitapide, using a Medication Adherence Scale for patients participating in the prospective phase.
  Unit of Measure: Medication Adherence Scale scores.

CONTACTS AND LOCATIONS:
Locations (30):
- France (5):
  - CHRU Lille - Centre Hospitalier Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire de Lyon (CHU Lyon), Lyon
  - Hôpital La Timone - Assistance Publique Hôpitaux de Marseille (AP-HM), Marseille
  - Hôpital La Pitié Salpêtrière - Groupe Hospitalier "La Pitié Salpêtrière - Charles Foix", Paris
  - Strasbourg University Hospital (CHU Strasbourg), Strasbourg
- Greece (3):
  - University General Hospital of Ioannina, Ioannina
  - University Hospital of Ioannina, Ioannina
  - METROPOLITAN HOSPITAL, Piraeus, Piraeus
- Italy (16):
  - Policlinico di Catanzaro - A.O.U. Mater Domini, Catanzaro, Calabria
  - Ospedale Sant'Anna e San Sebastiano, Caserta, Campania
  - Ospedale Monaldi - AORN dei Colli, Napoli, Napoli, Campania
  - Policlinico Federico II di Napoli, Napoli, Campania
  - Policlinico Sant'Orsola - Università di Bologna, Bologna, Emilia-Romagna
  - Arcispedale Sant'Anna - Università degli Studi di Ferrara, Ferrara, Emilia-Romagna
  - Ospedale Civile di Baggiovara - A.O.U. di Modena, Modena, Emilia-Romagna
  - DIMI - Dipartimento di Medicina Interna, Università di Genova, Genova, GE
  - Policlinico Umberto I - Sapienza Università di Roma, Rome, Lazio
  - Ospedale Bassini - ASST Nord Milano, Milan, Lombardy
  - Policlinico Paolo Giaccone - Università degli Studi di Palermo, Palermo, Sicily
  - Ospedale San Luigi Gonzaga, Orbassano, Torino
  - A.O.U. Città della Salute e della Scienza di Torino - Ospedale Molinette, Torino, Torino
  - CNR Gabriele Monasterio - Centro di Aferesi, Pisa, Pisa, Tuscany
  - Policlinico di Padova - A.O.U. di Padova, Padua, Veneto
  - Ospedale Borgo Trento - A.O.U. Integrata Verona, Verona, Veneto
- Netherlands (2):
  - Radboud University Medical Centre, Nijmegen
  - Rotterdam Erasmus Medical Center, Rotterdam
- United Kingdom (4):
  - Queen Elizabeth Hospital Birmingham (QEII - Birmingham), Birmingham, England
  - Harefield Hospital - Royal Brompton & Harefield NHS Foundation Trust, Harefield, England
  - Hammersmith Hospital - Imperial College Healthcare NHS Trust, London, England
  - Manchester University Hospital - NHS Foundation Trust, Manchester, England

IPD SHARING:
Plan to Share IPD: No
The LILITH study collects observational data on patients treated with lomitapide in compliance with data protection regulations (GDPR) and Good Clinical Practice (GCP) guidelines. At this time, individual participant data (IPD) sharing is not planned to ensure confidentiality and adherence to ethical and legal requirements. However, aggregated study results will be made available through scientific publications and regulatory reports.